CLINICAL TRIAL: NCT06380140
Title: Relationship Between Acute Phase Markers and Post-operative Pain in Open Tension-free Inguinal Hernia Repair: An Observational Study
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Augusto Lauro, Associate professor, University of Roma La Sapienza
Other Study IDs: cami3zgmxf3vqyc30ndmdqh6gfjid1
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Pain; Inguinal Hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing Open Tension-free Inguinal Hernia Repair
  Interventions: Procedure: Open Tension-free Inguinal Hernia Repair

INTERVENTIONS:
Procedure: Open Tension-free Inguinal Hernia Repair — A blood sample is taken the day after surgery

SUMMARY:
Many patients undergoing inguinal hernia repair are prone to developing acute and chronic post-operative pain.

The aim of the study is to show a possible correlation between pain and acute phase proteins in order to:

* predict the severity of pain;
* select most suitable pain relief therapy for the patient.

DETAILED DESCRIPTION:
The day after surgery, some serum markers are determined by a blood sample.

The markers analyzed are:

* Leukocytes;
* C-reactive protein (CRP);
* D-dimer;
* Fibrinogen;
* Neutrophil-to-Lymphocyte Ratio (NLR).

Pain level is assessed using the NRS scale at different times:

* 1st post-operative day;
* 7th post-operative day;
* One month after surgery;
* Three months after surgery;
* Six months after surgery.

Other data collected for the study are: gender, age, BMI.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing Open Tension-free Inguinal Hernia Repair

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes patients undergoing Open Tension-free Inguinal Hernia Repair
Sampling Method: Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship Between Post-operative Pain and C Reactive Protein (CRP) in Open Tension-free Inguinal Hernia Repair | one day
  The study compares post-operative pain, measured with the NRS scale, with CRP (μg/L) levels 24 hours after surgery
Relationship Between Post-operative Pain and D-dimer in Open Tension-free Inguinal Hernia Repair | one day
  The study compares post-operative pain, measured with the NRS scale, with D-dimer (μg/L FEU) levels 24 hours after surgery
Relationship Between Post-operative Pain and Fibrinogen in Open Tension-free Inguinal Hernia Repair | one day
  The study compares post-operative pain, measured with the NRS scale, with fibrinogen (g/L) levels 24 hours after surgery
Relationship Between Post-operative Pain and white blood cell count in Open Tension-free Inguinal Hernia Repair | one day
  The study compares post-operative pain, measured with the NRS scale, with white blood cell count (x 10^9/L) 24 hours after surgery
Relationship Between Post-operative Pain and Neutrophil to Lymphocyte Ratio (NLR) in Open Tension-free Inguinal Hernia Repair | one day
  The study compares post-operative pain, measured with the NRS scale, with Neutrophil to Lymphocyte Ratio (NLR) 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Augusto Lauro, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill AD, Banwell PE, Darzi A, Menzies-Gow N, Monson JR, Guillou PJ. Inflammatory markers following laparoscopic and open hernia repair. Surg Endosc. 1995 Jun;9(6):695-8. doi: 10.1007/BF00187942. PMID 7482166
- [Background] Kokotovic D, Burcharth J, Helgstrand F, Gogenur I. Systemic inflammatory response after hernia repair: a systematic review. Langenbecks Arch Surg. 2017 Nov;402(7):1023-1037. doi: 10.1007/s00423-017-1618-1. Epub 2017 Aug 22. PMID 28831565
- [Background] Vats M, Pandey D, Saha S, Talwar N, Saurabh G, Andley M, Kumar A. Assessment of systemic inflammatory response after total extraperitoneal repair and Lichtenstein repair for inguinal hernia. Hernia. 2017 Feb;21(1):65-71. doi: 10.1007/s10029-016-1543-1. Epub 2016 Nov 12. PMID 27838831
- [Background] Choi HR, Song IA, Oh TK, Jeon YT. Perioperative C-reactive protein is associated with pain outcomes after major laparoscopic abdominal surgery: a retrospective analysis. J Pain Res. 2019 Mar 27;12:1041-1051. doi: 10.2147/JPR.S187249. eCollection 2019. PMID 31114292
- [Background] Tarasov DA, Lychagin AV, Yavorovkiy AG, Lipina MM, Tarasova IA. C-reactive protein as marker of post-operative analgesic quality after primary total knee arthroplasty. Int Orthop. 2020 Sep;44(9):1727-1735. doi: 10.1007/s00264-020-04551-8. Epub 2020 Apr 16. PMID 32300831
- [Background] Esme H, Kesli R, Apiliogullari B, Duran FM, Yoldas B. Effects of flurbiprofen on CRP, TNF-alpha, IL-6, and postoperative pain of thoracotomy. Int J Med Sci. 2011 Mar 10;8(3):216-21. doi: 10.7150/ijms.8.216. PMID 21448308
- [Background] Rathee A, Chaurasia MK, Singh MK, Singh V, Kaushal D. Relationship Between Pre- and Post-Operative C-Reactive Protein (CRP), Neutrophil-to-Lymphocyte Ratio (NLR), and Platelet-to-Lymphocyte Ratio (PLR) With Post-Operative Pain After Total Hip and Knee Arthroplasty: An Observational Study. Cureus. 2023 Aug 20;15(8):e43782. doi: 10.7759/cureus.43782. eCollection 2023 Aug. PMID 37731439
- [Background] Shu B, Xu F, Zheng X, Zhang Y, Liu Q, Li S, Chen J, Chen Y, Huang H, Duan G. Change in perioperative neutrophil-lymphocyte ratio as a potential predictive biomarker for chronic postsurgical pain and quality of life: an ambispective observational cohort study. Front Immunol. 2023 Apr 12;14:1177285. doi: 10.3389/fimmu.2023.1177285. eCollection 2023. PMID 37122722
- [Background] Gonzalez-Callejas C, Aparicio VA, De Teresa C, Nestares T. Association of Body Mass Index and Serum Markers of Tissue Damage with Postoperative Pain. The Role of Lactate Dehydrogenase for Postoperative Pain Prediction. Pain Med. 2020 Aug 1;21(8):1636-1643. doi: 10.1093/pm/pnz325. PMID 31845982

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT06380140/Prot_SAP_000.pdf